CLINICAL TRIAL: NCT06442761
Title: Sickle Cell Disease Stem Cell Mobilization and Apheresis Using Motixafortide
Brief Title: SCD Stem Cell Mobilization and Apheresis Using Motixafortide
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Ayrmid Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: SCDSTEMM
Record Dates: First submitted 2024-05-13; First posted 2024-06-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: Stem Cell Mobilization; Apheresis; Motixafortide
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment-Arm A-Single Dose (Experimental): Part A: Participants who enroll early will be assigned to Part A. Part A participants will get one dose of the study drug and one stem cell collection process.
  Interventions: Drug: Motixafortide
- Treatment-Arm B-Two Daily Doses (Experimental): Part B: Participants who enroll later in the study will be assigned to Part B. Part B participants will get two doses of the study drug and two stem cell collection processes over two days (one on each day).
  Interventions: Drug: Motixafortide

INTERVENTIONS:
Drug: Motixafortide — Given Subcutaneously (under the skin).
  Other Names: APHEXDA™

SUMMARY:
This study is being done to see if the study drug, motixafortide, is safe in participants with sickle cell disease (SCD). Investigators also want to see if the drug will help the body increase the number of stem cells that can be collected for possible future transplant use.

PRIMARY OBJECTIVE

* To characterize the safety and tolerability of motixafortide in participants with SCD as determined by the incidence of adverse events (AEs).

SECONDARY OBJECTIVES

* To characterize the efficacy of a single dose (Part A) or two doses (Part B) of motixafortide for hematopoietic stem cell (HSC) mobilization and apheresis collection in participants with SCD as determined by the yield of CD34+ cells (CD34+ cells/kg).
* To measure the mobilization effects of single-day (Part A) or daily dosing (Part B) dosing with motixafortide in the peripheral blood in participants with SCD as determined by peak peripheral blood CD34+ counts
* To recommend a phase 2 dosing strategy based on safety, efficacy, and mobilization effects

DETAILED DESCRIPTION:
This study is divided into 2 parts. Participants will be assigned to a part based on when they enroll. Early in the study, participants will be assigned to part A. Later in the study, participants will be assigned to part B. In both parts, participants will receive the study drug, motixafortide, by an injection under the skin. About 4 hours after the injection, stem cells will be collected. Participants will follow-up within 7-10 days after the study drug and stem cell collection. Study staff will contact participants about 30 (±3) days after the last drug dose administration. The follow up may be conducted in person if the participant is in clinic during that follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Participants with severe sickle cell disease (SCD) who are ≥18 years of age and willing to donate autologous hematopoietic stem cells (HSCs) for advancing future gene therapy for SCD after collection of back-up product. Severe SCD, for the purpose of this study, will be defined as participants who are receiving chronic transfusion therapy due to SCD related complications or are eligible for or currently enrolled on an allogeneic transplant protocol.
* Participant must have a documented diagnosis of SCD with documentation of SCD genotype by medical history
* Participants should either have a central line in place, be able to undergo apheresis without the necessity of the insertion of a central venous catheter, or agree to have a central line placed if IV access is inadequate.
* ECOG performance status/Karnofsky score/Lansky score >80
* White blood cell (WBC) count >3.0 x 10^9/L, absolute neutrophil count (ANC) >1.0 x 10^9/L, and platelet count >150 x 10^9/L, and hemoglobin >7.0 gm/dL
* Adequate renal function defined as serum/plasma creatinine < 1.5 mg/dL and an estimated glomerular filtration rate (eGFR) of at least 60 mL/min/1.73 m^2 based on the CKD-Epi equation or the St. Jude equation.
* Adequate liver function defined as direct bilirubin < 2.5 times the upper limit of normal range; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 times the upper limit of normal range.
* Participant's cardiac function (i.e., ejection fraction >40%) and pulmonary status (i.e., no evidence of pulmonary hypertension) within the last 6 months must be sufficient to undergo apheresis, as assessed by the Principal Investigator or an independent physician evaluating the participant. If an assessment has not been done within the last 6 months, an echocardiogram will be performed.
* Negative serologic tests for syphilis, hepatitis B and C, HIV, and HTLV-1/II
* Feasible manual or automated exchange transfusion plan to achieve hemoglobin S (HbS) near 30% within one week of mobilization
* Female participants of childbearing age should have a negative pregnancy test.
* Participants of childbearing potential should agree to use of a highly effective form of contraception during treatment and for at least 1 month after the last dose of motixafortide. Women of childbearing potential must agree to use 2 methods of effective contraception: One barrier method (e.g. diaphragm, or condom or sponge, each of which are to be combined with a spermicide) and one hormonal method, unless she uses a highly effective method. Highly effective methods of contraception include:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
  * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomised partner
  * Sexual abstinence.

Exclusion Criteria:

* Active and painful splenomegaly or splenomegaly (size greater than upper limit of normal on examination).
* Participant who, by medical history, requires rare donor registry RBC units for transfusion, or is unable to receive routine transfusion. Eligible study participants must have undergone prior work-up for the presence of red cell alloantibodies and confirmation of available compatible blood product support
* Known allergy to or contraindication for motixafortide administration, or medications routinely administered during apheresis
* Participant who has had a prior autologous or allogeneic transplantation, inclusive of gene therapy
* Active viral, bacterial, fungal, or parasitic infection.
* History of cancer, excluding squamous carcinoma of the skin and cervical carcinoma in situ.
* Participant who has received experimental therapy within 4 weeks prior to providing informed consent
* Poorly controlled diabetes mellitus, as assessed by the Investigator
* Concomitant treatment with alternative investigational agent unable to be held for 30 days
* Unwillingness to use a highly effective method of contraception for 1 month after motixafortide
* Pregnancy
* Inability or unwillingness of research participant or legal guardian/ representative to give written informed consent.
* Inability or unwillingness of research participant to hold hydroxyurea for 30 days prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of motixafortide in participants with sickle cell disease (SCD) as determined by the incidence of adverse events. | 0 - 30 days

SECONDARY OUTCOMES:
To determine the yield of CD34+ cells/kg after a single or daily dose of motixafortide in participants with SCD. | 1 - 2 days
To determine the mobilization effects as determined by peripheral blood CD34+ counts/uL after a single or daily dose of motixafortide in participants with SCD. | 1 - 2 days
To recommend a phase 2 dosing strategy of one or two doses motixafortide in participants with SCD based on the incidence of adverse events | through study completion, an average of 1 year
To recommend a phase 2 dosing strategy for timing of apheresis based on peripheral blood CD34+ counts/uL after motixafortide administration in participants with SCD | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Leonard, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols